CLINICAL TRIAL: NCT02272530
Title: Analysis of Proteome and Pathophysiological Characteristics of Human Blood Cells
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator Prof. Dr. Malte Kelm, Heinrich-Heine University, Duesseldorf
Other Study IDs: Proteome
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Red Blood Cell; Peripheral Blood Mononuclear Cell; Endothelial NO-synthase
Keywords: Endothelial NO-synthase; red blood cell; erythrocytes; Peripheral Blood Mononuclear Cell; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy: 100 healthy volunteers in age of 20-75 years
- Patients: 100 patients with stable coronary artery disease and accordingly endothelial dysfunction

SUMMARY:
The aim of this study is to investigate wether change in endothelial nitric oxid synthase of blood cells (erythrocytes and peripheral blood mononuclear cells (PBMC)) has an influence on development and progression of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* Patients: stable coronary artery disease with accordingly endothelial dysfunction

Exclusion Criteria:

* acute inflammation (CRP>0,5 mg/dl, leucocyte >11000/dl)
* malignant diseases
* acute or terminated kidney disease
* relevant heart failure (NYHA III-IV)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 healthy volunteers and 100 patient with stable coronary artery disease
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Blood examination | baseline
  Following parameters will be examined:
  * Blood count (red cells, white cells, platelets, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red blood cell distribution width (RDW), mean platelet volume (MPV) )
  * Creatinin
  * Urea
  * Glucose
  * Glycated hemoglobin (HbA1c)
  * Cholesterol
  * Triglyceride
  * C-reactive Protein
  * Apolipoprotein

SECONDARY OUTCOMES:
Protein expression | baseline
  Determination with western blot
Asymmetric dimethylarginine (ADMA) and Cytokine | baseline
  Determination with enzyme-linked immunosorbent assay (ELISA).
Microparticles | baseline
  Determination with ELISA and flow cytometry
Immunocytochemistry | baseline
Nitric oxid metabolite and proteins in blood plasma, red blood cells and peripheral blood mononuclear cells (PBMN) | baseline
  Determination with reductive chemiluminescence
Nitric oxid and reactive oxygen species | baseline
  Determination with fluorescence coloring in flow cytometry and fluorescence microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof. MD, Principal Investigator — Department of Cardiology, Pneumology and Angiology, University Hospital Duesseldorf
Locations (1):
- University Hospital Duesseldorf, Düsseldorf, Germany